CLINICAL TRIAL: NCT02035436
Title: Substudy of the NONSEDA Trial (NCT01967680): Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Me-chanical Ventilation - Effects on Cognitive Function
Brief Title: Non-sedation Versus Sedation With a Daily Wake-up Trial in Critically Ill Patients Receiving Me-chanical Ventilation - Effects on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palle Toft (Other)
Collaborators: Kolding Sygehus (Other); University of Southern Denmark (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Sponsor-Investigator, Palle Toft, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S-20130025c
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Delirium; Cognition Disorders
Keywords: Respiration, artificial; Critcal care
MeSH Terms: conditions — Delirium; Cognition Disorders; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-sedation (Experimental): Non-sedation supplemented with pain management during mechanical ventilation.
  Interventions: Other: Non-sedation
- Sedation (Active Comparator): Current gold standard: Sedation with a daily wake-up trial.
  Interventions: Other: Control: Sedation

INTERVENTIONS:
Other: Non-sedation — Patients are awake or have natural sleep during mechanical ventilation. Pain is treated with morphine iv.
  Arms: Non-sedation
Other: Control: Sedation — Continuous iv-sedation (propofol first 48 hours, from then midazolam) to Ramsey 3-4 with a daily wake up attempt, where sedation is stopped until patient is awake.
  Arms: Sedation

SUMMARY:
Through many years, the standard care has been to use continuous sedation of critically ill patients during mechanical ventilation. However, preliminary randomised clinical trials indicate that it is beneficial to reduce the sedation level in these patients. The NONSEDA trial is an investigator-initiated, randomised, clinical, parallel-group, multinational, superiority trial designed to include 700 patients from at least six ICUs in Denmark, Norway and Sweden, comparing no sedation with sedation and a daily wake-up trial during mechanical ventilation. This is a substudy of the NONSEDA trial, concerning 250 patients included at trialsite Kolding, Denmark. The aim of the substudy is to assess the effects of no sedation on delirium during admission and cognitive function after discharge from ICU.

Our hypothesis is that critically ill patients who are not sedated during mechanical ventilation will have better cognitive function after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Endotracheally intubated
* Expected time on ventilator > 24 hours
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Severe head trauma where therapeutic coma is indicated
* Therapeutic hypothermia where therapeutic coma is indicated
* Status epilepticus where therapeutic coma is indicated
* Patient has participated in the study before
* Patient is transferred from another ICU with length of stay > 48 hours
* Patient is comatose at admission
* PaO2/FiO2 ≤ 9, if sedation is necessary for oxygenation
* Patient does not speak Danish, swedish or norwegian at a reasonable level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 3 months after discharge from ICU
  Cognitive t-score, in percentage, difference between the two groups. The t-score for each patient will be diagnosed by the neuropsycologist at a personal interview and use of following tests:
  * Span of numbers
  * Coding test
  * Trailmaking A+B
  * Rey auditory verbal learning test (immediate, recall)
  * Rey-Ostherrieth complex figure test (immediate, recall, recognition)
  * Word finding test (S-word, animals)
  * Stroop test (congruent+incongruent)

SECONDARY OUTCOMES:
Attention/concentration | 3 months after discharge from ICU
  T-score in the two groups for the cognitive domaine attention/concentration
Learning/memory | 3 months after discharge from ICU
  t-score in the two groups for the cognitive domaine: learning/memory
Executive dysfunction | 3 months after discharge from ICU
  t-score in the two groups for the cognitive domaine: executive dysfunction
Mental pace | 3 months after discharge from ICU
  t-score in the two groups for the cognitive domaine: mental pace
Hypoactive delirium | 3 months after discharge from ICU
  Occurrence of hypoactive delirium (RASS ≤ 0, CAM-ICU positive) in each group related to cognitive function at follow up
Agitated delirium | 3 months after discharge from ICU
  Occurrence of agitated delirium (RASS ≥ +2, CAM-ICU positive) in each group related to cognitive function at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Helene Joergensen, MD, Principal Investigator — Lillebaelt Hospital, Kolding
Locations (1):
- Lillebaelt Hospital, Kolding, Intensive Care Unit, Kolding, Denmark

REFERENCES:
- [Derived] Nedergaard HK, Jensen HI, Stylsvig M, Lauridsen JT, Toft P. Non-sedation versus sedation with a daily wake-up trial in critically ill patients recieving mechanical ventilation - effects on long-term cognitive function: Study protocol for a randomized controlled trial, a substudy of the NONSEDA trial. Trials. 2016 Jun 1;17(1):269. doi: 10.1186/s13063-016-1390-5. PMID 27250658